CLINICAL TRIAL: NCT00797823
Title: A Comparison of Two Sensor-Augmented Glycemic Control Systems in Persons With Type 1 Diabetes Mellitus: Subcutaneous (SC) Insulin and Glucagon Delivery vs. SC Insulin Only
Brief Title: Sensor-Augmented Insulin Delivery: Insulin Plus Glucagon Versus Insulin Alone
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Legacy Health System (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, W. Kenneth Ward, Senior Scientist, Legacy Health System
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: IRB4311
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Results first posted 2011-09-26 (Estimated); Last update posted 2011-10-07 (Estimated); Status verified 2009-08

CONDITIONS: Type 1 Diabetes
Keywords: diabetes; pancreas; beta cell; glucagon; insulin; hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Insulin Resistance; Hypoglycemia | interventions — Insulin Aspart; Glucagon; Glucagon-Like Peptide 1; Saline Solution; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- Insulin + Placebo (Placebo Comparator): Glycemic control of subject participants was managed by the closed-loop system which delivered insulin and normal saline (instead of glucagon) as a placebo, based upon algorithm calculations.
  Interventions: Drug: Insulin, Asp(B28)-; Drug: Placebo
- Insulin + Glucagon (Active Comparator): Glycemic control of subject participants was managed by the system which delivered insulin and glucagon based upon algorithm calculations.
  Interventions: Drug: Insulin, Asp(B28)-; Drug: Glucagon
- Pilot Study (Experimental): Pilot studies designed to assess safety of the system. Includes 6 participants undergoing 7 studies.
  Interventions: Drug: Insulin, Asp(B28)-; Drug: Glucagon; Drug: Placebo

INTERVENTIONS:
Drug: Insulin, Asp(B28)- — Insulin dosing and frequency calculated by Fading Memory Proportional Derivative algorithm
  Other Names: Aspart insulin; Novolog
Drug: Glucagon — During incipient hypoglycemia, glucagon was given in an attempt to prevent overt hypoglycemia. Dosing and frequency was calculated by the Fading Memory Proportional Derivative algorithm
  Other Names: Glucagen
  Arms: Insulin + Glucagon; Pilot Study
Drug: Placebo — Saline solution 0.9%
  Other Names: Normal saline, NaCl 0.9%
  Arms: Insulin + Placebo; Pilot Study

SUMMARY:
This study aims to test an insulin and glucagon delivery algorithm designed to be used in conjunction with a continuous glucose monitoring system. This combined glucose sensing/hormone delivery approach is a step on the way to eventual development of an artificial (or automated) pancreas. The insulin and glucagon delivery algorithm is based on the difference between the current blood glucose and the target glucose (proportional error) and the rate of change in blood glucose (derivative error), both adjusted for the recent glucose history. This algorithm is called the Fading Memory Proportional-Derivative (FMPD) Algorithm. The principal investigator of this study has published previous research regarding the use of this algorithm and found it to be well-suited to control blood glucose in type 1 diabetic animals. The addition of glucagon was helpful; better glycemic control with fewer glucose excursions were observed when small intermittent infusions of subcutaneous glucagon were given during times of impending low blood sugar (Ward et al. 2008).

DETAILED DESCRIPTION:
The objective of the current human study is to compare glycemic control in persons with Type 1 Diabetes using the FMPD Insulin plus Glucagon Delivery Algorithm vs. the FMPD Insulin-Alone Algorithm. Subjects will undergo two 28-hour sensor-augmented glycemic control studies. Each subject will be fitted with two short term continuous glucose monitoring systems and two subcutaneous (SC) infusion catheters. These catheters will allow for SC delivery of insulin and glucagon (or insulin plus a glucagon placebo). The accuracy of the wire sensors will be verified every 10 minutes with a venous blood glucose test. For the first 4 hours, the insulin and glucagon delivery will be controlled by venous blood in order to assess and compare the accuracy of the two sensors, after which the more accurate sensor (if it remains accurate) will control the FMPD algorithm. The main outcomes of our study are time spent in the target range (70 - 180 mg/dl) and the percentage of studies requiring intervention due to hypoglycemia (glucose < 70 mg/dl). The accuracy of the sensors over the life of the study will also be evaluated.

The specific system used in this study of frequent blood testing and the use of two separate infusion pumps is not feasible for every day use for individuals with diabetes. However, if the glucose control algorithm (with or without the use of glucagon) provides effective blood glucose management over long time periods the calculation program may be integrated into a continuous blood glucose monitoring system with an insulin and glucagon pump.

ELIGIBILITY:
Inclusion Criteria:

* Age 21-65, history of Type 1 Diabetes Mellitus for > 3 months.
* Women:

  * For women of childbearing potential, a negative urine pregnancy test is required on the first day of the study prior to sensor insertion AND the subject must agree to use contraception prior to and during the study.
  * For menopausal women or those who have undergone surgical sterilization, no pregnancy test or contraception will be required.
* Willingness to attend all clinic visits and participate in two 28-hour studies or one 9-hour study.
* Hemoglobin A1C of 5.0-10%. (Values below 5.0 suggest a severe tendency towards hypoglycemia, and values above 10% suggest severely uncontrolled diabetes with risk for ketoacidosis.)
* Body mass index of 19-35.

Exclusion Criteria:

* Pregnancy, lactation or refusal to use contraception.
* Use of any investigational drug during the 30 days prior to screening.
* Enrollment or participation in any other research studies 30 days prior to and during the entirety of sensor insertion.
* Current alcohol abuse, substance abuse, or severe mental illness (as judged by the Principal Investigator (PI)).
* Any prior cerebrovascular accident or major permanent neurological damage such as aphasia, hemiparesis, or dementia.
* A history of cerebrovascular disease or cardiovascular disease regardless of the time since occurrence.
* Coronary artery disease (symptomatic or asymptomatic) as manifested by unstable angina, acute coronary syndrome, myocardial infarction or therapeutic coronary procedure (e.g., Percutaneous Transluminal Coronary Angioplasty (PTCA), stent placement, Coronary Artery By-pass Grafting (CABG)) within the prior 6 months.
* Any degree of heart failure (as defined by New York Heart Association)..
* Renal insufficiency (serum creatinine of > 2.5).
* Current foot or leg ulceration.
* Peripheral arterial disease with uncontrolled claudication.
* Active uncontrolled malignancy except basal cell or squamous cell skin cancers.
* Concurrent illness, other than diabetic mellitus, that is not controlled by a stable therapeutic regimen.
* Hemoglobin A1C of less than 5.0 or greater than 10%.
* A total bilirubin level above 1.5 mg/dl.
* Medications: Oral or parenteral corticosteroids (glucocorticoid therapy) are exclusions; topical corticosteroids are not.
* Any chronic immunosuppressive medication (such as cyclosporine, azathioprine, sirolimus, or tacrolimus).
* Visual impairment that would prevent reading the display of the Medtronic Guardian® Receiver.
* Physical impairment that would prevent using the buttons of the Medtronic Guardian® Receiver.
* Serum Alanine Transaminase (ALT) or Aspartate Transaminase (AST) ≥3x the upper limit of normal.
* Serum albumin level of < 3.2 g/dl.
* Severe anemia as defined by a hematocrit of < 28%.
* Severe serum electrolyte abnormality (sodium, potassium, carbon dioxide, chloride).
* Cardiac rhythm disturbance characterized by: 2nd or 3rd degree heart block, bradycardia of less than 50 bpm (exception of bradycardia in an aerobic athlete), tachycardia of greater than 100 bpm, or any arrhythmia judged by the investigator to be exclusionary.
* A history of Human Immunodeficiency Virus (HIV) infection.
* An active hepatitis infection.
* Known allergy to any type of insulin
* Insulin resistance requiring more than 200 units of insulin per day
* Known bleeding disorders or chronic usage of warfarin.
* Any known seizure disorder.
* Past history of pheochromocytoma or a family history of Multiple Endocrine Neoplasia (MEN) 2A, MEN 2B, neurofibromatosis, or von Hippel-Lindau disease.
* Hypoglycemic unawareness or chronic hypoglycemia.
* A severe hypoglycemic event which required hospitalization within the past two years.
* Adrenal insufficiency.
* Insulinoma.
* Use of both acetaminophen and ascorbic acid.
* Impaired mentation or psychiatric diagnoses
* Uncontrolled candidiasis.
* Any known allergy to glucagon.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-11; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William K. Ward, MD, Principal Investigator — Legacy Health System
Locations (1):
- Legacy Research, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Oregon Health and Science University (OHSU) outpatient clinics in Portland, Oregon.
Pre-assignment Details: A total of 22 studies in 14 subjects were performed. 6 subjects participated in 7 9-hour pilot studies, 6 with insulin and glucagon and 1 with insulin + placebo to assess the safety of the protocol. 8 subjects then underwent 2 interventional studies each for a total of 16 studies, one with insulin and placebo and one with insulin and glucagon.
Groups:
- Insulin + Glucagon -> Insulin + Placebo): This group consists of x participants initially randomized to the insulin plus glucagon (latter to prevent hypoglycemia) intervention for glycemic control of type 1 diabetes during the first period, then insulin plus placebo in the second period. The control system was comprised of glucose sensors, a computer algorithm, and actuator pumps in a circuit meant to automatically adjust insulin and glucagon infusion rates based on glucose values delivered to the algorithm (a closed-loop system, as it is meant to exclude human intervention).
- Insulin + Placebo -> Insulin + Glucagon: This group consists of x participants initially randomized to the insulin plus placebo intervention for glycemic control of type 1 diabetes during the first period, then insulin plus glucagon (latter to prevent hypoglycemia) in the second period. The control system was comprised of glucose sensors, a computer algorithm, and actuator pumps in a circuit meant to automatically adjust insulin and glucagon infusion rates based on glucose values delivered to the algorithm (a closed-loop system, as it is meant to exclude human intervention).
- Pilot: Pilot studies included 6 participants, one of whom underwent an insulin + glucagon and an insulin + placebo study, while 5 underwent only one insulin + glucagon study.
Period: Pilot Studies
Arm/Group | Insulin + Glucagon -> Insulin + Placebo) | Insulin + Placebo -> Insulin + Glucagon | Pilot
Started | 0 (Not involved in pilot studies) | 0 (Not involved in pilot studies) | 6
Completed | 0 | 0 | 6
Not Completed | 0 | 0 | 0
Period: First Period (Initial Randomization)
Arm/Group | Insulin + Glucagon -> Insulin + Placebo) | Insulin + Placebo -> Insulin + Glucagon | Pilot
Started | 4 | 4 | 0 (Pilot studies only performed during initial period.)
Completed | 3 | 4 | 0
Not Completed | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0
Period: Second Period (Crossover)
Arm/Group | Insulin + Glucagon -> Insulin + Placebo) | Insulin + Placebo -> Insulin + Glucagon | Pilot
Started | 3 | 4 | 0
Completed | 3 | 4 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insulin + Glucagon -> Insulin + Placebo) | Insulin + Placebo -> Insulin + Glucagon | Pilot | Total
Number analyzed (Participants) | 4 | 4 | 6 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 6 | 14
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.3 (10.5) | 39.8 (10.7) | 35.1 (17.4) | 36.7 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 3 | 7
  Male | 2 | 2 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 6 | 14

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Closed Loop Diabetes Control
Description: Effectiveness of closed loop diabetes control will be measured by mean glucose.
Time Frame: 1 year
Population: The number of participants for analysis was determined was per protocol.
Measure: Mean (Standard Error); unit: mg/dl
Groups:
- Placebo Comparator: Insulin Alone: No glucagon given during closed loop control-insulin only
- Active Comparator: Insulin Plus Glucagon: Insulin plus glucagon given (latter to prevent hypoglycemia) for closed loop control.
Arm/Group | Placebo Comparator: Insulin Alone | Active Comparator: Insulin Plus Glucagon
Number analyzed (Participants) | 8 | 13
mg/dl | 136.9 (5.0) | 149.5 (5.5)

2. Secondary Outcome: Percent of Time Venous Blood Glucose <70 mg/dl
Time Frame: 1 year
Measure: Mean (Standard Error); unit: percent of time
Arm/Group | Placebo Comparator: Insulin Alone | Active Comparator: Insulin Plus Glucagon
Number analyzed (Participants) | 8 | 13
percent of time | 2.8 (0.67) | 1.15 (0.41)

ADVERSE EVENTS:
Time Frame: Over 1 year for entire research period, and over the study period for each individual study.
Arm/Group | Insulin + Glucagon -> Insulin + Placebo) | Insulin + Placebo -> Insulin + Glucagon | Pilot
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 1/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Insulin + Glucagon -> Insulin + Placebo) (N=4) | Insulin + Placebo -> Insulin + Glucagon (N=4) | Pilot (N=6)
Severe Hypoglycemia (Endocrine disorders) | 4 (55) | 4 (67) | 1 (1) — Venous blood glucose < 60 mg/dl, requiring treatment with intravenous (IV) dextrose.
Nausea and vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Nausea reported by patient (+/- vomiting), related to glucagon administration.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No